CLINICAL TRIAL: NCT03138291
Title: Efficacy of Oral Appliances on Obstructive Sleep Apnea During Pregnancy
Acronym: OSApod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nelly Huynh, Professor, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OSApod
Record Dates: First submitted 2016-03-15; First posted 2017-05-03 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Sleep Apnea, Obstructive; Pregnancy Related
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somnodent (Experimental): SomnoDent is a custom-made oral appliance for the treatment of mild to moderate obstructive sleep apnea. SomnoDent is worn during sleep to provide Continuous Open Airway Therapy by moving the lower jaw slightly forward. This movement tightens the soft tissue and muscles of the upper airway, which prevents obstructive apneas while sleeping.
  Interventions: Device: Somnodent

INTERVENTIONS:
Device: Somnodent — Each pregnant women will be treat with a Somnodent

SUMMARY:
Issue: The prevalence and severity of sleep-disordered breathing increases during pregnancy due to weight gain, physiological and hormonal changes. These sleep breathing disorders have a negative impact on perinatal health for both the mother and the child.The optimal treatment of obstructive sleep apnea in pregnancy is unknown. Although CPAP therapy is often the treatment of choice, the mandibular advancement appliance would be an interesting alternative to solve the matter.

Objectives: The main objective of this pilot study is to evaluate the feasibility of mandibular advancement device to treat sleep apnea during the 2nd and 3rd trimesters of pregnancy. Secondary objectives will be tools to plan a future randomized controlled trial to determine the efficacy of this treatment.

DETAILED DESCRIPTION:
Study design : Intervention Pilot Study uncontrolled experimental cohort

Population: 32 pregnant women with sleep apnea with an apnea - hypopnea index ( AHI ) ≥ 10 events / hr .

Methodology: The mandibular advancement appliance will be used with the chip DentiTracs to measure adhesion. Participation in this project requires five visits to the research team, including 3 visits at home. Participants will be recruited and granted in obstetrics MUHC. The questionnaires will be filled (Epworth Sleepiness Scale, Pittsburgh sleep quality and functional (FOSQ)). A sleep recording (PSG type II) will be done at home to confirm the diagnosis. The recording equipment will be returned to the research team by mail. During the second visit (clinical orthodontics), dental impressions in alginate will be made. At the 3rd visit (clinical orthodontics), the mandibular advancement appliance will be adjusted and instructions will be given. A weekly phone call follow-up will be ensured during this period of adjustment of the appliance. The fourth visit (at home) will consist of a sleep recording to evaluate the effect of treatment. A questionnaire comfort / secondary effects will be administered. For patients who have started their participation during their second trimester, a sleep recording at home (4a visit) will be realized in Q3 to assess whether it is necessary to change the titration of the appliance. The 5th visit (orthodontic clinic) will be 3-6 months after delivery. Participants will fulfill all the mentioned questionnaires and make a sleep recording at home without the appliance. Replace the appliance in place if AHI> 10. During the 4th and 5th visits, anthropometric data (ie, weight), and objective adhesion will be taken

ELIGIBILITY:
INCLUSION CRITERIA

* Adult women (≥ 18 years old)
* Pregnant women (between14 and 34 weeks)
* Sleep apnea with respiratory disturbance index (RDI) ≥ 5 events/hour
* Snoring or sleep apnea testimony by chamber partner

EXCLUSION CRITERIA

* Severe sleep apnea
* Evidence of a respiratory sleep disorder other than sleep apnea
* Body mass index greater than 40
* Use of medication that could affect breathing or sleep
* Abnormalities of the upper airway (oversized amygdala)
* Severe temporomandibular disorder
* Periodontal problems and untreated caries
* Poor dental hygiene
* Possible retention of OAM (Not enough teeth to retain the OAM in the mouth )

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
obstructive sleep apnea | 9 months
  Apnea hypopnea index

SECONDARY OUTCOMES:
adherence | 9 months
  A mini-recorder will be use to see how many hours a day the patient wear the appliance.

CONTACTS AND LOCATIONS:
Overall Officials: Sushmita Pamidi, MD, Principal Investigator — McGill University
Locations (1):
- University of Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Smocot J, Huynh N, Panyarath P, Kimoff RJ, Meltzer S, Drouin-Gagne L, Newbold R, Hebert C, Benedetti A, Arcache JP, Morency AM, Garfield N, Rey E, Pamidi S. Patterns of adherence to continuous positive airway pressure and mandibular advancement splints in pregnant individuals with sleep-disordered breathing. Sleep Breath. 2025 Apr 4;29(2):148. doi: 10.1007/s11325-025-03284-5. PMID 40183988
- [Derived] Huynh N, Drouin-Gagne L, Gilbert C, Arcache JP, Rompre P, Morency AM, Gagnon R, Kimoff J, Pamidi S. Adherence and efficacy of mandibular advancement splint treatment of sleep-disordered breathing during pregnancy: a pilot study. Sleep Breath. 2023 Jun;27(3):869-877. doi: 10.1007/s11325-022-02681-4. Epub 2022 Jul 13. PMID 35829947